CLINICAL TRIAL: NCT07239479
Title: Efficacy and Safety of Dexmedetomidine Combined With Desflurane in Laparoscopic Colectomy: A Randomized Double-Blind Controlled Clinical Trial (DEXDES Trial)
Brief Title: DEXDES Trial: Dexmedetomidine-Desflurane Combination in Laparoscopic Colectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tam Anh Research Institute (Other)
Collaborators: Tam Anh TP. Ho Chi Minh General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TA2.25.11
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Neoplasms
Keywords: Dexmedetomidine; Desflurane; General anesthesia; Colorectal surgery; ERAS; Hemodynamic stability
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Dexmedetomidine; Desflurane; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Arm 1 - Dexmedetomidine + Desflurane (Intervention Group):
  Dexmedetomidine bolus 1 µg/kg IV over 15 minutes before induction, followed by continuous infusion 0.5 µg/kg/h during surgery.
  Desflurane administered at 1 MAC with EtControl mode.
  Interventions: Drug: Dexmedetomidine + Desflurane
- Control Group (Placebo Comparator): Arm 2 - Desflurane + Normal Saline (Control Group):
  Normal saline infusion with identical timing and volume as the intervention group.
  Desflurane administered at 1 MAC with EtControl mode
  Interventions: Drug: Desflurane + Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine + Desflurane — Dexmedetomidine bolus 1 µg/kg IV over 15 minutes before induction, followed by continuous infusion 0.5 µg/kg/h during surgery.
  Desflurane administered at 1 MAC with EtControl mode.
  Arms: Intervention Group
Drug: Desflurane + Normal Saline — Normal saline infusion with identical timing and volume as the intervention group.
  Desflurane administered at 1 MAC with EtControl mode.
  Arms: Control Group

SUMMARY:
This randomized double-blind controlled clinical trial aims to evaluate the efficacy and safety of combining Dexmedetomidine with Desflurane in patients undergoing elective laparoscopic colectomy. The study will assess whether the combination can reduce Desflurane consumption, improve intraoperative hemodynamic stability, and enhance postoperative recovery compared to Desflurane alone.

DETAILED DESCRIPTION:
Dexmedetomidine, a selective alpha-2 adrenergic agonist, has sedative and analgesic properties without significant respiratory depression. Desflurane, a volatile anesthetic with low blood-gas solubility, allows rapid induction and emergence. Combining these two agents may provide anesthetic-sparing effects and promote faster postoperative recovery under ERAS protocols. This study will enroll 40 adult patients undergoing elective laparoscopic colectomy at Tam Anh General Hospital, Vietnam. Participants will be randomized into two groups: Dexmedetomidine + Desflurane versus Desflurane alone. The primary outcome is average Desflurane consumption per hour, with secondary outcomes including hemodynamic parameters, Fentanyl use, emergence quality, and incidence of postoperative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* ASA Physical Status I-II
* Elective laparoscopic colectomy
* Written informed consent provided

Exclusion Criteria:

* Severe cardiac, hepatic, or renal disease
* COPD or bronchial asthma
* Chronic opioid or psychotropic medication use
* Atrioventricular block (grade II-III), sick sinus syndrome
* Significant intraoperative bleeding or hemodynamic instability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Average Desflurane consumption per hour (mL/h) during surgery. | During surgery
  Average Desflurane consumption per hour (mL/h) during surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Tam Anh TP. Ho Chi Minh General Hospital, Ho Chi Minh City, Ho Chi Minh, Vietnam

IPD SHARING:
Plan to Share IPD: No
Individual patient data (IPD) will remain confidential. Aggregated, de-identified data may be shared upon reasonable request after study completion for academic purposes.